CLINICAL TRIAL: NCT04372342
Title: The Effect of Analgesic Drugs on Respiratory Center
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chun Pan (Other)
Collaborators: Southeast University, China (Other)
Responsible Party: Sponsor-Investigator, Chun Pan, Director, Southeast University, China
Organization: Southeast University, China (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: nalbuphine
Record Dates: First submitted 2020-01-21; First posted 2020-05-04 (Actual); Last update posted 2020-05-04 (Actual); Status verified 2020-04

CONDITIONS: The Effect of Analgesic Drugs on Respiratory Center
MeSH Terms: interventions — Nalbuphine; Remifentanil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nalbuphine (Experimental)
  Interventions: Drug: nalbuphine
- remifentanil (Placebo Comparator)
  Interventions: Drug: remifentanil

INTERVENTIONS:
Drug: nalbuphine — Nalbuphine hydrochloride has strong analgesic effect, quick effect and long time by stimulating receptor, and has partial antagonistic effect on the receptor, so the incidence of respiratory depression is low in theory.
  Other Names: remifentanil
  Arms: nalbuphine
Drug: remifentanil — remifentanil
  Arms: remifentanil

SUMMARY:
Opioids are commonly used in analgesic treatment of severe patients. Opioid receptors are divided into five types:,,, and.1 receptor is associated with analgesia and sedation above the spinal cord, while 2 receptor is associated with respiratory depression, bradycardia, euphoric sensation, pruritus, pupil contraction, inhibition of intestinal motility and other side effects.Κ receptors play a role of spinal analgesia, sedation and diuresis.Δ receptors associated with spinal analgesia and respiratory inhibition and regulate the activity of mu receptor.

Different opioid analgesics have different binding degree with different receptors, which determines the difference of analgesic effect and side effect, especially respiratory central inhibitory effect.Remifentanil is a pure opioid receptor agonist, mainly ACTS on the first and second receptors, binding to the second receptor is weak, in the analgesic, sedative effect, with opioid respiratory depression and hypotensive side effects, respiratory depression is dose dependent.Nalbuphine hydrochloride has strong analgesic effect, quick effect and long time by stimulating receptor, and has partial antagonistic effect on the receptor, so the incidence of respiratory depression is low in theory.The metabolic pathways of different opioids are also different. In particular, severe patients often need continuous opioid infusion for analgesia, which may lead to the accumulation of drugs and further affect the respiratory center.In the process of continuous application of different types of opioids to the analgesia of severe patients, the presence of respiratory center inhibition, the degree of inhibition and the dose-effect relationship have not been quantitatively evaluated.

ELIGIBILITY:
Inclusion Criteria:

Patients with tracheal intubation transferred to ICU after surgery;Stop the use of sedative drugs continue to pump more than 2h into the vein, anesthesia awake can cooperate with the command action;Can withstand PSV ventilation; need pain relief treatment

Exclusion Criteria:

Patients who cannot place transnasal gastric tube (EAdi catheter) beside the bed due to various reasons (such as massive gastrointestinal bleeding, esophagus and stomach surgery within the past 1 month, severe coagulation dysfunction);Patients with neuromuscular diseases: diseases that directly or indirectly inhibit respiratory centers and affect respiratory muscles;The patient is expected to die within 24 hours;Pregnant women, patients with malignant tumors;Patients with craniocerebral injury or ARDS who require deep sedation;Patients with agitated delirium.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-01-28 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Richmond Agitation-Sedation Scale | 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongda Hospital, Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No